CLINICAL TRIAL: NCT03424564
Title: A Single and Multiple Dose Pharmacokinetic Study of Perampanel in Chinese Healthy Subjects
Brief Title: Pharmacokinetic Study of Perampanel in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: E2007-C086-052
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-06

CONDITIONS: Healthy Subjects
Keywords: Perampanel; Pharmacokinetics; E2007; Chinese
MeSH Terms: interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Perampanel single-dose Part: 2 mg group (Experimental): Participants will receive a single 2 milligrams (mg) dose of perampanel orally under fasted conditions.
  Interventions: Drug: Perampanel
- Perampanel single-dose Part: 4 mg group (Experimental): Participants will receive a single 4 mg dose of perampanel orally under fasted conditions.
  Interventions: Drug: Perampanel
- Perampanel single-dose Part: 8 mg group (Experimental): Participants will receive a single 8 mg dose of perampanel orally under fasted conditions.
  Interventions: Drug: Perampanel
- Perampanel multiple-dose Part (Experimental): Participants will receive multiple oral dose of perampanel (2 milligrams per day [mg/day] from Day 1 to Day 7 and 4 mg/day from Day 8 to Day 21). Fasted condition is required for Days 1 and 21.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Oral Tablet
  Other Names: E2007

SUMMARY:
This study will be conducted to evaluate the pharmacokinetics of perampanel following single and multiple oral doses in Chinese healthy male and female participants.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in this study:

* Chinese healthy adult volunteers (males and females)
* Non-smoking, male or female age ≥18 years and ≤45 years old at the time of obtaining written consent. To be considered non-smokers, participants must have discontinued smoking from screening before first dosing.
* Participants with a Body Mass Index ≥18.5 and <24.5 kilograms per meters squared at screening
* Participants who undergo screening within 3 weeks before study treatment and are confirmed to be eligible by the investigator

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from this study:

* Participants who weigh less than 50 kilograms
* Females who are breastfeeding or pregnant at Screening or Baseline
* Females of childbearing potential
* Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks before first dosing
* Evidence of disease that may influence the outcome of the study within 4 weeks before first dosing
* Any history of gastrointestinal surgery that may affect pharmacokinetic profiles of perampanel at Screening
* Any clinically abnormal symptom or organ impairment found by medical history at Screening, and physical examinations, vital signs, electrocardiogram (ECG) finding, or laboratory test results that require medical treatment at Screening
* A prolonged QT/corrected QT (QTc) interval (QTc interval for heart rate using Fredericia's formula >450 milliseconds) as demonstrated by a repeated ECG at Screening or Baseline

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Single-dose Part: Mean value of the maximum observed concentration (Cmax) postdose of perampanel | 0-336 hours postdose
Single-dose Part: Mean value for the time at which the highest drug concentration occurs (tmax) postdose of perampanel | 0-336 hours postdose
Single-dose Part: Mean value for area under the concentration-time curve from zero time to 24 hours (AUC[0-24h]) postdose of perampanel | 0-24 hours postdose
Single-dose Part: Mean value for area under the concentration-time curve from zero time to time of last quantifiable concentration (AUC[0-t]) postdose of perampanel | 0-336 hours postdose
Single-dose Part: Mean value for area under the concentration-time curve from zero time extrapolated to infinite time (AUC[0-inf]) postdose of perampanel | 0-336 hours postdose
Single-dose Part: Mean value for the terminal phase rate constant (λz) postdose of perampanel | 0-336 hours postdose
Single-dose Part: Mean value for terminal elimination phase half-life (t1/2) postdose of perampanel | 0-336 hours postdose
Single-dose Part: Mean value for apparent total clearance following oral administration (CL/F) postdose of perampanel | 0-336 hours postdose
Single-dose Part: Mean value for the apparent volume of distribution at terminal phase (Vz/F) postdose of perampanel | 0-336 hours postdose
Single-dose Part: Mean residence time (MRT) postdose of perampanel | 0-336 hours postdose
Multiple-dose Part: Mean value of Cmax postdose of perampanel on Day 1 | 0-24 hours postdose on Day 1
Multiple-dose Part: Mean minimum observed concentration (Cmin) postdose of perampanel on Day 1 | 0-24 hours postdose on Day 1
Multiple-dose Part: Mean tmax postdose of perampanel on Day 1 | 0-24 hours postdose on Day 1
Multiple-dose Part: Mean AUC(0-24h) postdose of perampanel on Day 1 | 0-24 hours postdose on Day 1
Multiple-dose Part: Mean value of area under the concentration-time curve over the dosing interval on multiple dosing (AUC[0-τ]) | 0-24 hours postdose of perampanel on Day 21
Multiple-dose Part: Mean value of the average steady-state concentration (Css,av) postdose of perampanel on Day 21 | 0-24 hours postdose on Day 21
Multiple-dose Part: Mean value of the maximum observed concentration at steady state (Css,max) postdose of perampanel on Day 21 | 0-24 hours postdose on Day 21
Multiple-dose Part: Mean value of the minimum observed concentration at steady state (Css,min) postdose of perampanel on Day 21 | 0-24 hours postdose on Day 21
Multiple-dose Part: Mean value of peak-trough fluctuation (PTF) postdose of perampanel on Day 21 | 0-24 hours postdose on Day 21
Multiple-dose Part: Mean time at which the highest drug concentration occurs at steady state (tss,max) postdose of perampanel on Day 21 | 0-24 hours postdose on Day 21
Multiple-dose Part: Mean time at which the lowest drug concentration between dosing intervals occurs at steady state (tss,min) postdose of perampanel on Day 21 | 0-24 hours postdose on Day 21
Multiple-dose Part: Mean value of t1/2 postdose of perampanel on Day 21 | 0-336 hours postdose on Day 21
Multiple-dose Part: Mean value of apparent total clearance following oral administration at steady state (CLss/F) postdose of perampanel on Day 21 | 0-24 hours postdose on Day 21
Multiple-dose Part: Mean value of Vz/F postdose of perampanel on Day 21 | 0-336 hours postdose on Day 21
Multiple-dose Part: Mean value of the accumulation ratio | 0-24 hours postdose of perampanel on Days 1 and 21

CONTACTS AND LOCATIONS:
Locations (1):
- Eisai Trial Site, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Jing S, Shiba S, Morita M, Yasuda S, Lin Y. A Single- and Multiple-Dose Pharmacokinetic Study of Oral Perampanel in Healthy Chinese Subjects. Clin Drug Investig. 2023 Mar;43(3):155-165. doi: 10.1007/s40261-022-01241-8. Epub 2023 Feb 6. PMID 36746851